CLINICAL TRIAL: NCT00394693
Title: Phase II Clinical Trial of Intra-lesional Administration of TG1042 (Adenovirus-Interferon-gamma) in Patients With Relapsing Primary Cutaneous B-Cell Lymphomas.
Brief Title: Study to Evaluate the Safety and Efficacy of Adeno-IFN Gamma in Cutaneous B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG1042.06
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma, B-Cell
Keywords: Primary CBCL including (WHO/EORTC classification 2005); Primary cutaneous marginal zone B-cell lymphoma; Primary cutaneous follicle center B-cell lymphoma; Primary cutaneous diffuse large B-cell other than leg type; Histologically consistent with primary CBCL; Relapse or active disease
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

INTERVENTIONS:
Genetic: Adenovirus Interferon gamma — intra-tumoral injections, 1 dose per lesion, up to 6 simultaneous lesions.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a four-month dosing period of intra-lesional injection of TG1042 in patients with relapsing CBCL.

Patients will receive intra-tumoral injections of an adenoviral vector construct containing the human interferon gamma gene (TG1042), in an attempt to enhance immune responses with anti-tumor activity. This local administration induces tumour cell killing at the injected tumour sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy all the following criteria for entry into the protocol:

Primary CBCL including (according to WHO/EORTC classification 2005) :

* Primary cutaneous marginal zone B-cell lymphoma
* Primary cutaneous follicle center B-cell lymphoma
* Primary cutaneous diffuse large B-cell other than leg type

  * Histologically consistent with primary CBCL.
  * Relapse or active disease after radiotherapy or other adequate therapy if radiotherapy was contra-indicated (chemotherapy, surgical excision, interferonα, rituximab).
  * Performance status of 0, 1 on the Eastern Cooperative Oncology Group (ECOG) scale (See Appendix E).
  * Minimum Life Expectancy > 3 months.
  * Adequate blood count: hemoglobin >= 10.0 g/dL; White Blood Count (WBC) >= 3.0 x 109/L; and platelet count >= 75 x 109/L.
  * Adequate hepatic function: bilirubin =< 1.5 times the upper limit of normal and serum transaminase (SGOT and SGPT)=< 2.5 times the upper limit of normal.
  * Adequate renal function: creatinine =< 1.5 times the upper limit of normal.
  * Written informed consent from patient.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Primary cutaneous diffuse large B-cell lymphoma, leg type.
* Primary cutaneous intravascular large B-cell lymphoma.
* Extracutaneous involvement (sign of B-cell lymphoma on thoraco-abdominal CT scan and/or PET scan and/or on bone marrow biopsy).
* No histologic documentation of CBCL.
* History of known Human Immuno-deficiency Virus, Human Hepatitis B or C positive serology or other active systemic infections.
* Serious uncontrolled, concomitant medical disorders.
* Concomitant therapy for CBCL: surgical resection, radiotherapy, corticosteroid, chemotherapy, rituximab…(not limited listing)
* Major surgery in previous 4 weeks preceding the 1st injection.
* Pregnancy at study entry or who become pregnant during the study or women who are breast feeding.
* Males and females of reproductive potential who refuse to use adequate protection against pregnancy (intra-uterine device, hormonal contraception or diaphragm/condom and spermicide) during the conduct of the study and for three months after the last injection.
* Participation in another experimental protocol during the study period and within 4 weeks prior to the first injection.
* Patient previously included in this study.
* Non compliance with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Regression and disappearance of lesions | end of cycle
Safety | visit

SECONDARY OUTCOMES:
Quality of Life | visit

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Northwestern University Medical School, Chicago, Illinois
  - M.D. Anderson Cancer Center, Houston, Texas
- France (2):
  - Hopital Lapeyronie, Montpellier
  - Hopital de l'Hotel-Dieu, Nantes
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Dreno B, Urosevic-Maiwald M, Kim Y, Guitart J, Duvic M, Dereure O, Khammari A, Knol AC, Derbij A, Lusky M, Didillon I, Santoni AM, Acres B, Bataille V, Chenard MP, Bleuzen P, Limacher JM, Dummer R. TG1042 (Adenovirus-interferon-gamma) in primary cutaneous B-cell lymphomas: a phase II clinical trial. PLoS One. 2014 Feb 24;9(2):e83670. doi: 10.1371/journal.pone.0083670. eCollection 2014. PMID 24586226
- [Derived] Accart N, Urosevic-Maiwald M, Dummer R, Bataille V, Kehrer N, Niculescu C, Limacher JM, Chenard MP, Bonnefoy JY, Rooke R. Lymphocytic infiltration in the cutaneous lymphoma microenvironment after injection of TG1042. J Transl Med. 2013 Sep 25;11:226. doi: 10.1186/1479-5876-11-226. PMID 24063735
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/lymphoma.html